CLINICAL TRIAL: NCT01862757
Title: Pilot Study of Strength Testing in Overweight Women With or Without Insulin Resistance
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130130; 13-H-0130
Record Dates: First submitted 2013-05-23; First posted 2013-05-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-03-13

CONDITIONS: Obesity
Keywords: Obesity; Insulin; Skeletal Muscle; Strength Testing
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Some people who are obese may have decreased muscle strength. They may have greater muscle mass shown in scans, but they show poor results in exercise tests. Poor muscle strength might cause some of the difficulty with exercise performance. Researchers want to test muscle strength in the arms and legs of overweight women. They will also see how insulin resistance affects muscle strength in these women.

Objectives:

* To test muscle strength in overweight women.
* To see if insulin resistance affects muscle strength.

Eligibility:

- Women at least 18 years of age who are overweight (body mass index greater than 25 kg/m2).

Design:

* Participants will be asked to fast before having an initial blood test to measure glucose and insulin levels.
* On a different day, they will have the strength testing. The first test will measure leg muscle strength by testing the quadriceps and the hamstrings. The second test will measure arm muscle strength by testing the biceps and triceps. The final test will measure hand muscle (grip) strength.
* All the tests should take about an hour.

DETAILED DESCRIPTION:
We have observed in our protocol (08-H-0108: Effects of Worksite Wellness Interventions on Vascular Function, Insulin Sensitivity and High-Density Lipoprotein in Overweight or Obese Women) that despite increased lean (muscle) mass in the extremities as measured by dual x-ray absorptiometry, obese women have poorer exercise tolerance than overweight women who have less muscle mass.1 Exercise testing, however, is an integrated function of cardiopulmonary capacity, in addition to muscle strength and endurance. We propose to determine whether muscle strength of elbow flexors and knee extensor muscle groups correlates with muscle mass of these groups in overweight and obese women selected for normal or abnormal insulin sensitivity. Our hypothesis is that subjects with impaired insulin sensitivity and high insulin levels will have greater muscle mass but lower muscle strength than subjects with normal insulin sensitivity and normal insulin levels. This is a feasibility study to be conducted in 10 non-diabetic women (5 with insulin resistance, 5 with normal insulin sensitivity) who previously participated in 08-H-0108, the outcome of which will provide data for planning a larger study of muscle mass and strength which may be important to achieving exercise goals important to successful weight loss.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Non-diabetic female employees of NIH who participated in protocol 08-H-0108 and underwent insulin sensitivity testing and also protocol 02-H-0050 for muscle mass determination.
* BP< 140/90 mmHg (medications allowed)
* Subject understands protocol and provides written, informed consent.

EXCLUSION CRITERIA:

* Medical or surgical condition that would prohibit upper and lower extremity strength testing (e.g., painful arthritis, prior knee or elbow surgery)
* Infection or injury to hand, knee or elbow requiring medical attention within 3 months of testing

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05-06; Primary Completion 2013-06-14 (Actual); Study Completion 2015-03-13 (Actual)

PRIMARY OUTCOMES:
To determine whether increased extremity muscle mass associated with obesity, diminished insulin sensitivity and high insulin levels is associated with diminished strength. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Richard O Cannon, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Leon B, Jenkins S, Pepin K, Chaudhry H, Smith K, Zalos G, Miller BV 3rd, Chen KY, Remaley AT, Waclawiw MA, Sumner AE, Cannon RO 3rd. Insulin and extremity muscle mass in overweight and obese women. Int J Obes (Lond). 2013 Dec;37(12):1560-4. doi: 10.1038/ijo.2013.45. Epub 2013 Mar 28. PMID 23609936
- [Background] Park SW, Goodpaster BH, Strotmeyer ES, de Rekeneire N, Harris TB, Schwartz AV, Tylavsky FA, Newman AB. Decreased muscle strength and quality in older adults with type 2 diabetes: the health, aging, and body composition study. Diabetes. 2006 Jun;55(6):1813-8. doi: 10.2337/db05-1183. PMID 16731847
- [Background] Kimball SR, Farrell PA, Jefferson LS. Invited Review: Role of insulin in translational control of protein synthesis in skeletal muscle by amino acids or exercise. J Appl Physiol (1985). 2002 Sep;93(3):1168-80. doi: 10.1152/japplphysiol.00221.2002. PMID 12183515